CLINICAL TRIAL: NCT02808182
Title: Postprandial Fatty Acid Metabolism in the Natural History of Type 2 Diabetes (T2D): Relative Contribution of Dietary vs Systemic Fatty Acids to Lean Tissue Fatty Acid Fluxes and Oxidative vs Non-oxidative Pathways
Brief Title: Postprandial Fatty Acid Metabolism in the Natural History of Type 2 Diabetes (T2D)
Acronym: AGL11
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, André Carpentier, Tenured Professor, Université de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2016-1196
Record Dates: First submitted 2016-04-14; First posted 2016-06-21 (Estimated); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Impaired Glucose Tolerance
MeSH Terms: conditions — Glucose Intolerance | interventions — Niacin; Biopsy

ARMS (4):
- A0: PET/scan with [11C] palmitate (Other): A bolus of 180 MBq of [11C]-acetate at time 90min and PET acquisition
  Interventions: Procedure: Biopsy; Other: liquid meal
- A1: PET/scan with [11C] palmitate (Other): A bolus injection of 180 MBq of [11C]-acetate at time 90min, followed by PET acquisition
  Interventions: Drug: Nicotinic acid; Procedure: Biopsy; Other: liquid meal
- B0: PET/scan with [18F]-FTHA (Other): At time 0, a standard liquid meal will be drunk over 20 minutes with 70 MBq of 18FTHA . PET acquisition at time 90 min.
  Interventions: Other: [7,7,8,8-2H]-palmitate; Other: [U-13C]-palmitate; Other: liquid meal
- B1: PET/scan with [18F]-FTHA (Other): At time 0, a standard liquid meal will be drunk over 20 minutes with 70 MBq of 18FTHA followed by a PET acquisition at time 90 min.
  Interventions: Drug: Nicotinic acid; Other: [7,7,8,8-2H]-palmitate; Other: [U-13C]-palmitate; Other: liquid meal

INTERVENTIONS:
Drug: Nicotinic acid — oral administration of nicotinic acid (100mg at 0, 30, 60, 90, 120, 180, 240 and 300 min) to minimize WAT intracellular lipolysis
  Other Names: Niacin
  Arms: A1: PET/scan with [11C] palmitate; B1: PET/scan with [18F]-FTHA
Other: [7,7,8,8-2H]-palmitate — using i.v. administration of [7,7,8,8-2H]-palmitate (in 25% human albumin) from time -60 to +360 min
  Arms: B0: PET/scan with [18F]-FTHA; B1: PET/scan with [18F]-FTHA
Other: [U-13C]-palmitate — oral administration of [U-13C]-palmitate (0.2 g mixed into the liquid meal) at time 0 min
  Arms: B0: PET/scan with [18F]-FTHA; B1: PET/scan with [18F]-FTHA
Procedure: Biopsy — A subcutaneous abdominal 0.5-g adipose tissue biopsy will be performed at the end of protocols A0 and A1
  Arms: A0: PET/scan with [11C] palmitate; A1: PET/scan with [11C] palmitate
Other: liquid meal — At time 0, a standard liquid meal (400 mL, 906 kcal, 33g-fat/34g-protein/101g-carbohydrates i.e. 33%/17%/50% calories) will be drunk over 20 minutes

SUMMARY:
Lipotoxicity-causing fatty acid overexposure and accretion in lean tissues leads to insulin resistance and impaired pancreatic β-cell function - the hallmarks of T2D - contributing to associated complications such as heart failure, kidney failure and microvascular diseases. Proper dietary fatty acid (DFA) storage in white adipose tissue (WAT) is now thought to prevent lean-tissue lipotoxicity. Using novel Positron-Emission Tomography (PET) and stable isotopic tracer methods which were developed in Sherbrooke, the investigator showed that WAT storage of DFA is impaired in people with pre-diabetes or T2D. The investigator also showed that this impairment is associated with greater cardiac DFA uptake, as well as subclinical left-ventricular systolic and diastolic dysfunction. Then, It has been found that modest weight loss in pre-diabetics, after a one-year lifestyle intervention, improved WAT DFA storage, curbed cardiac DFA uptake, and restored associated left-ventricular dysfunction. It has been also found that a 7-day low-saturated fat, low-calorie diet raised insulin sensitivity but did not restore WAT or cardiac DFA metabolism. Whether WAT DFA storage directly impacts cardiac DFA uptake is not known. Importantly, the investigator recently uncovered marked sex-specific differences in WAT DFA metabolism. These may explain, at least in part, sex-related differences in the cardiac DFA uptake, which occurs in pre-diabetes. Higher spillover of WAT DFA into circulating Non-Esterified Fatty Acid (NEFA) appears to be linked in women to greater cardiac DFA uptake, as opposed to direct cardiac chylomicron triglycerides (TG) uptake in men. Here, the investigator will isolate and compare organ-specific fatty acid uptake occurring postprandially from chylomicron-TG vs. NEFA pools, as well as the oxidative vs. non-oxidative intracellular metabolic pathways associated with increased cardiac DFA uptake in pre-diabetic men and women.

ELIGIBILITY:
Inclusion Criteria:

* For healthy subjects: fasting glucose < 5.6, 2-hour post 75g Oral Glucose Tolerance Test (OGTT) glucose < 7.8 mmol/l and HbA1c < 5.8%
* For subject with glucose intolerance (IGT): 2-hour post 75g OGTT glucose at 7.8-11.1 mmol/l on two separate occasions and HbA1c of 6.0 to 6.4%

Exclusion Criteria:

* overt cardiovascular disease as assessed by medical history, physical exam, and abnormal ECG
* treatment with a fibrate, thiazolidinedione, beta-blocker or other drug known to affect lipid or carbohydrate metabolism (except statins, metformin, and other antihypertensive agents that can be safely interrupted)
* presence of liver or renal disease, uncontrolled thyroid disorder, previous pancreatitis, bleeding disorder, or other major illness
* smoking (>1 cigarette/day) and/or consumption of >2 alcoholic beverages per day
* prior history or current fasting plasma cholesterol level > 7 mmol/l or fasting TG > 6 mmol/l
* any other contraindication to temporarily interrupt current meds for lipids or hypertension
* being pregnant
* not be barren

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-01-17 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2021-05 (Actual)

PRIMARY OUTCOMES:
Plasma NEFA appearance rate | 2 years
  NEFA appearance will be measured using i.v. administration of [7,7,8,8-2H]-palmitate (in 25% human albumin) from time -60 to +360 min, as slightly modified from previous descriptions, using Steele's non steady-state equations. Blood samples to measure plasma palmitate, oleate, linoleate, and total NEFA levels, [7,7,8,8-2H]-palmitate enrichments by GC/MS-MS.
Cardiac and hepatic uptake | 2 years
  will be determined using 11C-palmitate PET/CT. 180 MBq will be administered by bolus injection at postprandial time 90min. After a transmission scan and regional CT (40mA), a 30-min dynamic list-mode PET acquisition will be performed starting at time 90 min on a 18 cm-high thoraco-abdominal segment to include the left cardiac ventricle and most of the liver on a Philips Gemini TOF PET/CT
WAT spillover NEFA appearance rates | 2 years
  WAT spillover NEFA will be determined from oral administration of [U-13C]-palmitate.
  Blood samples to measure plasma [U-13C]-palmitate and chylomicron-TG [U-13C]-palmitate enrichment by GC/MS-MS
oxidative metabolism of NEFA | 2 years
  will be assessed by using 13C-palmitate
cardiac and hepatic DFA uptake | 2 years
  will be assessed using PET/CT method with oral administration of 18FTHA
whole-body organ-specific DFA partitioning | 2 years
  will be determined by whole-body CT (16 mA) followed by PET acquisition of 18FTHA

SECONDARY OUTCOMES:
Insulin sensitivity | 2 years
  will be determined using the HOMA-IR (based on fasting insulin and glucose levels)
Insulin secretion rate | 2 years
  will be assessed using deconvolution of plasma C-peptide with standard C-peptide kinetic parameters
β-cell function | 2 years
  will be assessed by calculation of the disposition index (DI) that is insulin secretion in response to the ambient insulin
WAT size | 2 years
  by biopsy fixed in formalin
hormonal response | 2 years
  will be determined using a multiplex assay system
Lipoprotein lipase activity | 2 years
  will be assessed as on frozen 150-mg portions from biopsy

CONTACTS AND LOCATIONS:
Locations (1):
- centre de recherche du CHUS, Sherbrooke, Quebec, Canada

REFERENCES:
- [Derived] Montastier E, Ye RZ, Noll C, Amrani M, Frisch F, Fortin M, Bouffard L, Phoenix S, Sarrhini O, Cunnane SC, Guerin B, Turcotte EE, Carpentier AC. Nicotinic acid increases adipose tissue dietary fatty acid trapping and reduces postprandial hepatic and cardiac fatty acid uptake in prediabetes. Eur J Pharmacol. 2025 Jul 5;998:177563. doi: 10.1016/j.ejphar.2025.177563. Epub 2025 Mar 27. PMID 40157702
- [Derived] Ye RZ, Montastier E, Noll C, Frisch F, Fortin M, Bouffard L, Phoenix S, Guerin B, Turcotte EE, Carpentier AC. Total Postprandial Hepatic Nonesterified and Dietary Fatty Acid Uptake Is Increased and Insufficiently Curbed by Adipose Tissue Fatty Acid Trapping in Prediabetes With Overweight. Diabetes. 2022 Sep 1;71(9):1891-1901. doi: 10.2337/db21-1097. PMID 35748318
- [Derived] Montastier E, Ye RZ, Noll C, Bouffard L, Fortin M, Frisch F, Phoenix S, Guerin B, Turcotte EE, Lewis GF, Carpentier AC. Increased postprandial nonesterified fatty acid efflux from adipose tissue in prediabetes is offset by enhanced dietary fatty acid adipose trapping. Am J Physiol Endocrinol Metab. 2021 Jun 1;320(6):E1093-E1106. doi: 10.1152/ajpendo.00619.2020. Epub 2021 Apr 19. PMID 33870714
- See also: Total Postprandial Hepatic Nonesterified and Dietary Fatty Acid Uptake Is Increased and Insufficiently Curbed by Adipose Tissue Fatty Acid Trapping in Prediabetes With Overweight — https://pubmed.ncbi.nlm.nih.gov/35748318/
- See also: Increased postprandial nonesterified fatty acid efflux from adipose tissue in prediabetes is offset by enhanced dietary fatty acid adipose trapping — https://pubmed.ncbi.nlm.nih.gov/33870714/